CLINICAL TRIAL: NCT01046422
Title: A Double-blind, Placebo-Controlled, Parallel-group, Randomized, Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of BMS-770767 in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Either Diet and Exercise Alone or on a Background of Metformin
Brief Title: Safety Study of BMS-770767 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB117-003; 2009-014308-79 (EudraCT Number)
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — BMS-770767; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- BMS-770767 ± metformin (Treatment A) (Experimental)
  Interventions: Drug: BMS-770767; Drug: Metformin
- BMS-770767 ± metformin (Treatment B) (Experimental)
  Interventions: Drug: BMS-770767; Drug: Metformin
- BMS-770767 ± metformin (Treatment C) (Experimental)
  Interventions: Drug: BMS-770767; Drug: Metformin
- BMS-770767 ± metformin (Treatment D) (Experimental)
  Interventions: Drug: BMS-770767; Drug: Metformin
- Placebo ± metformin (Treatment E) (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: BMS-770767 — Capsule, Oral, 15mg, Active, Daily, 28 days
  Arms: BMS-770767 ± metformin (Treatment A)
Drug: BMS-770767 — Capsule, Oral, 50mg, Active, Daily, 28 days
  Arms: BMS-770767 ± metformin (Treatment B)
Drug: BMS-770767 — Capsule, Oral, 150mg, Active, Daily, 28 days
  Arms: BMS-770767 ± metformin (Treatment C)
Drug: BMS-770767 — Capsule, Oral, 50mg BID, Active, Daily, 28 days
  Arms: BMS-770767 ± metformin (Treatment D)
Drug: Placebo — Capsule, Oral, 0mg, Daily, 28 days
  Arms: Placebo ± metformin (Treatment E)
Drug: Metformin — Tablet, Oral, ≥ 1500mg, Active, Daily, 28 days

SUMMARY:
The purpose of this study is to determine if BMS-770767 is safe, well tolerated, measure its levels in the blood (pharmacokinetics), and measure the levels of chemicals (biomarkers) that may be affected by this drug (pharmacodynamics) in a type 2 diabetes patient population

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes with inadequate glycemic control and treated with either diet and exercise alone, or with stable doses (≥ 1500mg/d) of metformin for at least 8 weeks prior to screening
* HbA1c ≥ 7.0% and ≤ 10.0% with FPG ≤ 240mg/dL (13.3 mmol/dL)

Exclusion Criteria:

* Women of childbearing potential
* History of diabetic ketoacidosis or hyperosmolar nonketotic coma
* Significant cardiovascular history
* History of unstable or rapidly progressing renal disease
* Impaired renal function defined by a serum creatinine > 1.4mg/dL (124 µmol/L) for women and >1.5mg/dL (133 µmol/L) for men
* Active liver disease and /or significant abnormal liver function defined as AST > 3X ULN and/or ALT > 3XULN and /or serum total bilirubin > 2.0mg/dl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Fasting Plasma Glucose Improvement | Within seven days following dosing

SECONDARY OUTCOMES:
Mean daily glucose (3-day 7 pt-fingerstick) | Within 28 days following dosing
Four (4)-hour post-prandial glucose AUC | Within 28 days following dosing
HbA1C | Within 28 days following dosing
Lipid profiles | Within 28 days following dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- United States (2):
  - Marina Raikhel, Md, Lomita, California
  - Nevada Alliance Against Diabetes, Las Vegas, Nevada
- Australia (5):
  - Local Institution, Caboolture, Queensland
  - Local Institution, Meadowbrook, Queensland
  - Local Institution, Daw Park, South Australia
  - Local Institution, Geelong, Victoria
  - Local Institution, Nedlands, Western Australia
- Canada (9):
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Mount Pearl, Newfoundland and Labrador
  - Local Institution, Brampton, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Charlottetown, Prince Edward Island
  - Local Institution, Drummondville, Quebec
  - Local Institution, Lachine, Quebec
  - Local Institution, Laval, Quebec
  - Local Institution, Montreal, Quebec
- South Korea (2):
  - Local Institution, Incheon
  - Local Institution, Suwon

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx